CLINICAL TRIAL: NCT04963920
Title: A Prospective, Randomized, Multicenter, Single-blind, Controlled Study to Assess the Performance of the Cytosorb® 300 ml Device for Shock Reversal in Patients With Vasoplegic Septic Shock
Brief Title: A RCT to Assess the Performance of CytoSorb for Shock Reversal in Patients With Vasoplegic Septic Shock
Acronym: PROCYSS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment for the study is currently on hold to allow for a protocol amendment. This revision aims to align the study design with changes in clinical practice since the trial's initiation.
Sponsor: CytoSorbents Europe GmbH (Industry)
Collaborators: BRAHMS GmbH (Unknown); MedInnovation GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S18
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SoC+CytoSorb treatment (Experimental): patients allocated to this group, will receive CytoSorb therapy in addition to the standard of care therapy according to applicable guidelines
  Interventions: Device: Cytosorb® 300 ml
- Standard of Care (SoC) (No Intervention): patients allocated to this group will receive only standard of care therapy according to applicable guidelines

INTERVENTIONS:
Device: Cytosorb® 300 ml — patients will receive CytoSorb therapy in addition to standard of care therapy according to applicable guidelines
  Arms: SoC+CytoSorb treatment

SUMMARY:
To assess the performance of the CytoSorb® 300 mL device for shock reversal in patients with vasoplegic septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with standard of care (SOC) according to guidelines for sepsis/septic shock for > 6 and < 30 hours prior to randomization
2. Vasoplegic septic shock*, requiring NA ≥ 0.2 µg/kg/min at the time of randomization, despite adequate fluid resuscitation to maintain MAP ≥ 65 mmHg after at least 6 hours of guideline-oriented initial therapy, including continuous NA administration
3. Lactate >2 mmol/l and <8 mmol/l at baseline
4. IL-6 ≥ 1000 ng/l at screening
5. Minimum 18 years of age
6. Provide voluntary consent to participate in the study either directly or via a legally authorized representative (LAR) or in accordance to the procedure after determination of an emergency situation according to Art. 68 (1) MDR, as applicable

   * (Septic shock is defined according to the SCCM / EISCM task force Sepsis-3 definition [Singer 2016])

Exclusion Criteria:

1. Patients with an abdominal source of infection without a source control intervention at the time of randomization OR a planned additional surgical intervention within the first 28 hours after randomization
2. Administration of any other vasopressors than NA at time of randomization and within the first 28 hours after randomization
3. Indication for va-ECMO at baseline OR a planned va-ECMO within the first 28 hours after randomization
4. Patients with a steroid therapy above Cushing-threshold dose (e.g. 30 mg hydrocortisone/d or 6 mg prednisolone/d) for more than 30 days prior to baseline
5. Cytokine-specific antibody therapy before inclusion
6. Anticipated interruption of CytoSorb® therapy for more than 2 hours within the first 26 hours after start of intervention
7. Conditions with a poor 90-day chance of survival because of an uncorrectable medical condition such as poorly controlled neoplasm, or other moribund end-stage disease states in which death was perceived to be imminent
8. Cancer patients currently on chemotherapy with cytostatics, tyrosine kinase inhibitors, or a treatment with antibodies (e.g. PD-1-inhibitors)
9. Acute traumatic brain injury
10. Decision to limit or withdraw treatment within the study and/or observation period in the ICU
11. Pregnancy / breast feeding
12. Participation in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage change in noradrenaline (NA) dose 24 hours after baseline, assessed as mean over the time window 22 to 26 hours after baseline | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, Prof, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf (UKE)
Locations (18):
- Germany (18):
  - Department of Intensive Care Medicine, University Medical-Center Hamburg-Eppendorf, Hamburg, Hamburg
  - Department of Nephrology and Medical Intensive Care, Charité - University Medical Center, Berlin
  - Department of Anesthesiology and Operative Intensive Care Medicine (CBF), Charité - Universitätsmedizin Berlin, Berlin
  - Department of Anesthesiology and Critical Care Medicine, University Hospital of Dresden, Dresden
  - Klinikum Emden, Emden
  - Clinic for Interdisciplinary Intensive Care and Intermediate Care, HELIOS Hospital Erfurt, Erfurt
  - Department of Nephrology, University Hospital Essen, Essen
  - Department of Anesthesiology, Intensive-Care Medicine and Pain Therapy, University Hospital Frankfurt, Frankfurt am Main
  - Department of Anesthesiology, Emergency and Intensive Care Medicine, University of Göttingen, Göttingen
  - Department of Internal Medicine B, Cardiology, Pneumology, Infectious Diseases, Intensive Care Medicine, University Hospital Greifswald, Greifswald
  - Department of Anesthesiology, Surgical Intensive Care, Emergency and Pain Medicine, Ruhr- University Bochum, Klinikum Herford, Herford, Germany, Herford
  - Department of Anaesthesiology, Intensive Care and Pain Therapy, Saarland University Medical Center and Saarland University Faculty of Medicine, Homburg
  - Department of Anesthesiology, Operative Intensive Care Medicine, Pain Management and Emergency Medicine, Hospital Ibbenbüren, Ibbenbueren
  - Department of Internal Medicine, Neurology and Dermatology, Interdisciplinary Internal Intensive Care Medicine, University Leipzig, Leipzig
  - Department of Internal Medicine II, Technical University of Munich, Munich
  - Department of Anaesthesiology and Intensive Care Medicine, Technical University of Munich, Munich
  - Center for Emergency and Intensive Care Medicine, Hospital Ernst von Bergmann, Potsdam
  - Department of Anesthesiology and Intensive Care Medicine, Rostock University Medical Centre, Rostock

IPD SHARING:
Plan to Share IPD: No